CLINICAL TRIAL: NCT05992545
Title: Diabetes Care Via a Mobile Application on Integrating Physical and Mental Health: A Pilot Study
Brief Title: Mobile Application for Integrative Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Bae, Jae Hyun, Clinical Associate Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DangDangCare
Record Dates: First submitted 2023-07-23; First posted 2023-08-15 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 2; Depression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile application 'DangDang Care' under usual care (Experimental): The intervention group receives 'DangDang Care' alongside usual diabetes care.
  Interventions: Device: Mobile application 'DangDang Care' under usual care
- Usual care (No Intervention): The control group receives only usual diabetes care.

INTERVENTIONS:
Device: Mobile application 'DangDang Care' under usual care — The application incorporates a behavioral activation program to provide psychological support and enhance diabetes self-management for people with type 2 diabetes experiencing depressive symptoms, alongside conventional medical therapy.
  The intervention group receives the mobile application with usual care.
  Other Names: DangDang Care
  Arms: Mobile application 'DangDang Care' under usual care

SUMMARY:
The investigators have developed a mobile application named 'DangDang Care' (which conveys the meaning of managing diabetes confidently and consistently through psychological care) designed to provide psychological support and enhance diabetes self-management for people with type 2 diabetes experiencing depressive symptoms. The application incorporates a behavioral activation program. Subsequently, the investigators conducted a 12-week randomized controlled trial, enrolling individuals with type 2 diabetes and mild-to-moderate depression, with the assistance of public health centers. The trial aimed to assess the effectiveness and feasibility of the application in promoting consistent diabetes management through added psychological care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 to 80 years with type 2 diabetes
* Individuals belonging to disadvantaged populations, such as medical aid beneficiaries or those classified as low-income groups
* Mild-to-moderate depressive symptoms, defined as a Patient Health Questionnaire-9 (PHQ-9) score between 5 and 19
* Capable of reading and understanding Korean and using a mobile application
* Having a clear understanding of the study's purpose and providing written consent

Exclusion Criteria:

* Type 1 diabetes or gestational diabetes
* Diabetes complications that hindered diabetes self-management
* Severe depressive symptoms that made app usage and completion of the self-report questionnaire difficult
* Serious mental illnesses other than depressive symptoms (e.g., schizophrenia and related disorders, bipolar and related disorders, or neurodegenerative disorders)
* Serious life-threatening medical conditions
* Physical conditions that impeded mobility
* A history of traumatic brain injury
* Unwillingness to complete the questionnaire and provide personal information

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Changes in Patient Health Questionnaire-9 (PHQ-9) scores | By week 12
  The PHQ-9 is a 9-item self-report scale developed to assess the presence and severity of depression within the past 2 weeks. It was adapted for use with Korean participants. Respondents rate how often they have been bothered by each problem on a 4-point Likert scale ranging from 0 to 3. The total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms, and a cutoff score of 10 is used.
Changes in Generalized Anxiety Disorder-7 (GAD-7) scores | By week 12
  The GAD-7 is a brief self-report scale that assesses generalized anxiety disorder, comprising 7 items. Respondents rate the frequency of experiencing symptoms related to generalized anxiety disorder over the past 2 weeks using a 4-point Likert scale ranging from 0 to 3. Total scores range from 0 to 21, with higher scores indicating more severe anxiety. In this study, we used the Korean version of the GAD-7, accessible on the Patient Health Questionnaire website.
Changes in Korean version of the Perceived Stress Scale (K-PSS) scores | By week 12
  The Perceived Stress Scale (PSS), originally developed in 1983, was translated into Korean in 2010 and 2012. The K-PSS consists of 10 items, and respondents rate their responses on a 5-point Likert scale ranging from 0 to 4. The total score ranges from 0 to 40, with higher scores indicating higher perceived stress levels.
Changes in Brief Diabetes Distress Screening Instrument (DDS-2) scores | By week 12
  The DDS-2 is a brief version of the Diabetes Distress Scale, developed in 2008, and was translated into Korean in 2020. It consists of 2 items, and each item assesses the emotional burden of diabetes and the stress of diabetes management and treatment on a 6-point Likert scale ranging from 1 to 6. The total score ranges from 2 to 12, with higher scores indicating higher levels of diabetes-related stress.
Changes in European Quality of Life-5 Dimensions 3 Level (EQ-5D-3L) index | By week 12
  The EQ-5D-3L is a tool developed by the Euro Quality of Life Group to assess health-related quality of life. It comprises a descriptive system with five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents rate their current health state within each domain using three levels. The evaluative system included the EQ-5D-3L index. We employed the EQ-5D-3L index to calculate utility values for health states and evaluate the overall quality of life.
Changes in Diabetes Self-Efficacy Scale (DSES) scores | By week 12
  The DSES, originally developed by the Stanford Patient Education Research Center in 2009, was used in its Korean version translated by Young Sun Yeom in her thesis in 2010. It comprises 8 items, and respondents rate their level of confidence in successfully performing self-care behaviors on a 10-point Likert scale ranging from 1 to 10. Higher scores indicate a higher level of self-efficacy in managing diabetes.
Changes in Diabetes Care Profile-Social Support Scale (DCP-SSS) scores | By week 12
  The Diabetes Care Profile (DCP), developed in 1996, measures psychosocial factors and diabetes treatment. For this study, only the instrumental and emotional support subscales were utilized, and they were translated into Korean in 2007. The scale was modified to fit the study's purpose, resulting in a total of 9 items, excluding 3 items not relevant to the study. Each item was answered on a 5-point Likert scale from 1 to 5, with higher scores indicating higher perceived social support.
Changes in Diabetes Self-Management Behaviors for Older Koreans (DSMB-O) scores | By week 12
  The DSMB-O was developed in 2016 and is based on the self-management standards proposed by the American Association of Diabetes Educators, considering the characteristics of older adults with type 2 diabetes in Korea. The scale consists of a total of 14 questions, with 9 questions answered on a 4-point Likert scale from 0 to 3, and 5 dichotomous questions. The total score ranges from 0 to 30, with higher scores indicating higher levels of diabetes self-care behaviors.

SECONDARY OUTCOMES:
Changes in glycated hemoglobin (%) | By week 12
  Measures average blood glucose levels over the past 2-3 months through venous blood sampling.
Changes in fasting plasma glucose levels (mg/dL) | By week 12
  Measures glucose levels after an 8-hour fasting period through venous blood sampling.
Change in lipid profiles, including total cholesterol, triglycerides, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol (mg/dL) | By week 12
  Measures total cholesterol, triglycerides, high-density lipoprotein cholesterol (HDL-C), and low-density lipoprotein cholesterol (LDL-C) after an 8-hour fasting period through venous blood sampling.

OTHER OUTCOMES:
Persistent changes in Patient Health Questionnaire-9 (PHQ-9) scores | By week 16
  The PHQ-9 is a 9-item self-report scale developed to assess the presence and severity of depression within the past 2 weeks. It was adapted for use with Korean participants. Respondents rate how often they have been bothered by each problem on a 4-point Likert scale ranging from 0 to 3. The total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms, and a cutoff score of 10 is used.
Persistent changes in Generalized Anxiety Disorder-7 (GAD-7) scores | By week 16
  The GAD-7 is a brief self-report scale that assesses generalized anxiety disorder, comprising 7 items. Respondents rate the frequency of experiencing symptoms related to generalized anxiety disorder over the past 2 weeks using a 4-point Likert scale ranging from 0 to 3. Total scores range from 0 to 21, with higher scores indicating more severe anxiety. In this study, we used the Korean version of the GAD-7, accessible on the Patient Health Questionnaire website.
Persistent changes in Korean version of the Perceived Stress Scale (K-PSS) scores | By week 16
  The Perceived Stress Scale (PSS), originally developed in 1983, was translated into Korean in 2010 and 2012. The K-PSS consists of 10 items, and respondents rate their responses on a 5-point Likert scale ranging from 0 to 4. The total score ranges from 0 to 40, with higher scores indicating higher perceived stress levels.
Persistent changes in Brief Diabetes Distress Screening Instrument (DDS-2) scores | By week 16
  The DDS-2 is a brief version of the Diabetes Distress Scale, developed in 2008, and was translated into Korean in 2020. It consists of 2 items, and each item assesses the emotional burden of diabetes and the stress of diabetes management and treatment on a 6-point Likert scale ranging from 1 to 6. The total score ranges from 2 to 12, with higher scores indicating higher levels of diabetes-related stress.
Persistent changes in European Quality of Life-5 Dimensions 3 Level (EQ-5D-3L) index | By week 16
  The EQ-5D-3L is a tool developed by the Euro Quality of Life Group to assess health-related quality of life. It comprises a descriptive system with five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents rate their current health state within each domain using three levels. The evaluative system included the EQ-5D-3L index. We employed the EQ-5D-3L index to calculate utility values for health states and evaluate the overall quality of life.
Persistent changes in Diabetes Self-Efficacy Scale (DSES) scores | By week 16
  The DSES, originally developed by the Stanford Patient Education Research Center in 2009, was used in its Korean version translated by Young Sun Yeom in her thesis in 2010. It comprises 8 items, and respondents rate their level of confidence in successfully performing self-care behaviors on a 10-point Likert scale ranging from 1 to 10. Higher scores indicate a higher level of self-efficacy in managing diabetes.
Persisent changes in Diabetes Care Profile-Social Support Scale (DCP-SSS) scores | By week 16
  The Diabetes Care Profile (DCP), developed in 1996, measures psychosocial factors and diabetes treatment. For this study, only the instrumental and emotional support subscales were utilized, and they were translated into Korean in 2007. The scale was modified to fit the study's purpose, resulting in a total of 9 items, excluding 3 items not relevant to the study. Each item was answered on a 5-point Likert scale from 1 to 5, with higher scores indicating higher perceived social support.
Persistent changes in Diabetes Self-Management Behaviors for Older Koreans (DSMB-O) scores | By week 16
  The DSMB-O was developed in 2016 and is based on the self-management standards proposed by the American Association of Diabetes Educators, considering the characteristics of older adults with type 2 diabetes in Korea. The scale consists of a total of 14 questions, with 9 questions answered on a 4-point Likert scale from 0 to 3, and 5 dichotomous questions. The total score ranges from 0 to 30, with higher scores indicating higher levels of diabetes self-care behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No